CLINICAL TRIAL: NCT04327934
Title: Mechanisms of Hypertension in Women With Polycystic Ovary Syndrome
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unble to complete all arms of the planned study due to Covid stoppage and difficulty with recruiting and getting enrolled participants to return post Covid.
Sponsor: Yale University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000020950; R01HL135089-01A1 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2020-03-31 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Polycystic Ovary Syndrome; Hypertension
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hypertension | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; ganirelix; Methyltestosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Healthy Control (Active Comparator): Healthy control participants.
  Interventions: Drug: GnRH antagonist; Drug: GnRH antagonist + MethylTESTOSTERone 5 MG
- AE-PCOS (Experimental): Participants with AE-PCOS.
  Interventions: Drug: GnRH antagonist; Drug: GnRH antagonist + MethylTESTOSTERone 5 MG

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist up to 16 days.
  Other Names: Antagon
Drug: GnRH antagonist + MethylTESTOSTERone 5 MG — GnRH antagonist + MethylTESTOSTERone 5 MG up to 5 days.
  Other Names: Antagon + MethylTESTOSTERone

SUMMARY:
Women with androgen excess polycystic ovary syndrome (AE-PCOS) leads to hypertension.

DETAILED DESCRIPTION:
Our scientific premise is that in AE-PCOS women, the androgen-dominant hormonal milieu causes BP increases via sympathetic activation, vasoconstriction and renal sympathetic nervous system activation. Moreover, this androgen-dominant milieu increases BP via activation of the renin-angiotensin system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Polycystic Ovary Syndrome
* Able to inject study drug
* Able to swallow pills

Controls:

-Diagnosis of Insulin resistance

Exclusion Criteria:

* Any woman that does not fit the inclusion criteria
* Males

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Obese Insulin Resistant (IR) women
Enrollment: 28 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Stachenfeld, PhD, Principal Investigator — Yale University
Locations (1):
- The John B Pierce Laboratory, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We will recruit subjects using flyers, our clinics, and social media. Dates 12/01/2017 - 04/29/2022; We were not able to reach recruit goals because our laboratory closed during Covid. When we reopened, we lost a one interested subject, and found greater challenges to recruit subjects.
Period: Overall Study
Arm/Group | Healthy Control | AE-PCOS
Started | 14 | 14
Completed | 7 | 9
Not Completed | 7 | 5
Not completed — Did not qualify | 7 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for people that completed the study- which is defined as those that were allocated, began and completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | AE-PCOS | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6) | 24 (5) | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 5 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Baroreflex Response to LBNP
Description: forearm blood flow (ultrasound)/mean arterial pressure as a linear function of lower body negative pressure. This is an important measure of autonomic control of blood pressure. Indicating the the sensitivity of changes in vessel diameter in response to blood pooling (induced by lower body negative pressure).
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: Arbitrary Units/Beat/mmHg
Groups:
- Healthy Control: Healthy Control
  GnRH antagonist: GnRH antagonist up to 16 days.
  GnRH antagonist + MethylTESTOSTERone 5 MG: GnRH antagonist + MethylTESTOSTERone 5 MG up to 5 days.
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
Arbitrary Units/Beat/mmHg
  Baseline | 0.98 (1.35) | 1.36 (0.96)
  GnRH antagonist | 1.9 (3.0) | 4.28 (6.51)
  GnRH antagonist with GnRH + Testosterone | 0.68 (0.65) | 1.46 (0.76)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Equivalence — We compared groups across treatments; p = 0.018, ANOVA

2. Primary Outcome: Free Plasma Testosterone Levels
Description: Concentration of testosterone in blood.
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
mg/dL
  Baseline | 0.76 (0.57) | 2.72 (1.13)
  GnRH | 0.67 (0.39) | 1.06 (0.31)
  GnRH + Testosterone | 1.34 (0.23) | 2.19 (0.19)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Equivalence — We compared across groups and within groups over time; p < 0.016, ANOVA
Statistical Analysis 2: Comparison: Healthy Control; Test type: Equivalence — We compared across groups and within groups over time; p = 0.08, ANOVA

3. Primary Outcome: Renal Response to LBNP
Description: POST Lower body negative pressure Plasma renin activity
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: ng/mL ANG/hour
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
ng/mL ANG/hour
  Baseline | 1.05 (0.82) | 1.10 (0.46)
  GnRH | 0.54 (0.33) | 1.14 (1.31)
  GnRH+Testosterone | 0.83 (0.71) | 1.36 (1.51)

4. Primary Outcome: Renal Responses to LBNP
Description: PRE lower body negative pressure Plasma renin activity
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: ng/mL ANG/hour
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
ng/mL ANG/hour
  Baseline | 0.53 (0.48) | 0.85 (0.97)
  GnRH | 0.42 (0.21) | 0.79 (1.24)
  GnRH + Testosterone | 0.63 (0.43) | 0.76 (0.75)

5. Primary Outcome: Resting Systolic Blood Pressure
Description: Blood pressure prior to lower body negative pressure
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Population: Systolic Blood Pressure
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | AE-PCOS | Healthy Control
Number analyzed (Participants) | 9 | 7
mm Hg
  Baseline | 128 (15) | 123 (13)
  GnRH | 131 (10) | 124 (16)
  GnRH +Testosterone | 130 (12) | 121 (16)
Statistical Analysis 1: Comparison: AE-PCOS vs Healthy Control; Test type: Other; p = 0.05, Friedman's test — Friedman's tests to compare slopes

6. Primary Outcome: Final Systolic Blood Pressure
Description: SBP at the end of lower body negative pressure
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
mm Hg
  Baseline | 105 (21) | 99 (23)
  GnRH | 109 (16) | 113 (12)
  GnRH + Testosterone | 117 (16) | 121 (10)

7. Primary Outcome: Resting Sympathetic Activity
Description: Total sympathetic nerve activity
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: burst/100 heart beats
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
burst/100 heart beats
  Baseline | 14.4 (4.4) | 10.3 (2.0)
  GnRH | 7.9 (0.8) | 6.9 (1.5)
  GnRH + Testosterone | 13.4 (3.6) | 14.5 (5.0)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Other; p = 0.023, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Control vs AE-PCOS; Test type: Other; p < 0.04, ANOVA

8. Primary Outcome: Sympathetic Baroreflex
Description: microneurography, diastolic blood pressure (finipres) This is an important measure of autonomic control of blood pressure. Indicating the the sensitivity of changes in muscle sympathetic nerve activity in response to small changes in blood pressure induced by drug perfusion (modified Oxford).
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: Gain (bursts/100 heart beats/ mm Hg)
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
Gain (bursts/100 heart beats/ mm Hg)
  Baseline | -0.479 (0.085) | -0.496 (0.142)
  GnRH | -0.468 (0.101) | -0.640 (0.171)
  GnRH+Testosterone | -0.445 (0.087) | -0.487 (0.124)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Equivalence — We compared groups across treatments; p = 0.0023, ANOVA

9. Secondary Outcome: Aldosterone
Description: Plasma aldosterone concentration
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
pg/mL
  Baseline | 75.7 (41.4) | 136.5 (60.1)
  GnRH | 44.0 (37.0) | 127.8 (70.5)
  GnRH+testosterone | 46.1 (28.6) | 98.7 (46.6)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Other; p < 0.04, ANOVA

10. Secondary Outcome: Renal Responses
Description: P[ACE], angiotensin-converting enzyme
Time Frame: Baseline, assessed at 7 days of GnRH, assessed at 16 days GnRH+ 5 days of Testosterone
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Healthy Control | AE-PCOS
Number analyzed (Participants) | 7 | 9
µg/L
  Baseline | 38.2 (14.7) | 101.9 (93.4)
  GnRH | 43.4 (27.3) | 77.7 (76.5)
  GnRH + Testosterone | 40.6 (14.1) | 44.2 (43.2)
Statistical Analysis 1: Comparison: Healthy Control vs AE-PCOS; Test type: Other; p < 0.04, ANOVA

ADVERSE EVENTS:
Time Frame: Six to eight weeks
Description: One subject experienced mild back pain during LBNP. Another experienced an incident of lupus on an experimental day, not due to our studies. However this was reported to our IRB.
Arm/Group | Healthy Control | AE-PCOS
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Control (N=14) | AE-PCOS (N=14)
non serious adverse event (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
non serious adverse event (Immune system disorders) | 0 (0) | 1 — lupus flair unrelated to study

LIMITATIONS AND CAVEATS:
Our primary limitation was stoppage due to Covid (our laboratory was forced to close). We also had a very challenging time recruiting subjects when we reopened after the three-month closure under new rules. Subjects who had been enrolled did not return, and new subjects were difficult to recruit. Thus, we were not able to complete all arms of the planned study. We were able to answer our primary questions regarding autonomic function in women with PCOS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/34/NCT04327934/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT04327934/ICF_001.pdf